CLINICAL TRIAL: NCT05063695
Title: Pragmatic Study Comparing Outcomes of Multimodal Epidural and Erector Spinae Catheter Pain Protocols After Pectus Surgery
Brief Title: Pectus ESC Outcomes and Comparative Effectiveness Study
Acronym: PectusESC
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0374
Record Dates: First submitted 2021-09-17; First posted 2021-10-01 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Pectus Excavatum; Pain, Postoperative
MeSH Terms: conditions — Funnel Chest; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural: Patients who underwent Nuss procedure under epidural protocol (between January and December of 2019)
- ESP: Patients who underwent Nuss procedure using ESP catheter protocol (June 2020 to April 2021)
  Interventions: Other: Multimodal Erector spinae catheter protocol

INTERVENTIONS:
Other: Multimodal Erector spinae catheter protocol — Patients either received multimodal epidural or ESP protocol
  Other Names: Multimodal epidural protocol
  Groups: ESP

SUMMARY:
Investigators hypothesize that Erector spinae catheter pain management protocol would allow patients to have earlier and more effective rehabilitation with decreased length of hospital stay. The aims are to compare LOS between the two groups (epidural and ES groups). Secondary aims are to compare recovery outcomes (mobilization time), time required to do the blocks, pain scores and opioid use during hospitalization and on follow up after discharge until Pain clinic visit, side effects, family satisfaction and readmissions among the two groups. In addition, in-hospital and post-discharge outcomes in subjects who received ESP protocol will be studied.

DETAILED DESCRIPTION:
Retrospective study - Electronic medical records of consecutive patients who underwent pectus surgery between January and December of 2019 (epidural protocol) and those who underwent same procedure between June 2020 to May 2021, will be evaluated. Covariates and outcomes described in sections below will be recorded from EMR. The data included records from flowsheets, pain team notes based on follow up questionnaires administered by phone after discharge until after ESP catheters were removed, as well as pain clinic notes.

ELIGIBILITY:
Inclusion Criteria:

* Age>8 years
* Diagnosis of pectus excavatum who underwent Nuss procedure
* Pain regimen included either epidural catheter or ES catheters

Exclusion Criteria:

* Developmental delay
* prior pectus repair
* concomitant procedures

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with pectus excavatum who underwent Nuss procedure
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Upto 10 days after surgery
  Date of surgery to hospital discharge
Mobilization | After surgery in-hospital, phone calls until POD6, pain clinic and surgery clinic postop visit (within 4 weeks after surgery)
  Meeting PT goals

SECONDARY OUTCOMES:
Pain measures | After surgery in-hospital, phone calls until POD6, pain clinic and surgery clinic postop visit (within 4 weeks after surgery)
  Pain scores postoperative and opioid/benzodiazepine use
Side effects | After surgery in-hospital, phone calls until POD6, pain clinic and surgery clinic postop visit (within 4 weeks after surgery)
  ED visit, readmission, numbness, infection, LA toxicity etc.

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muhly WT, Beltran RJ, Bielsky A, Bryskin RB, Chinn C, Choudhry DK, Cucchiaro G, Fernandez A, Glover CD, Haile DT, Kost-Byerly S, Schnepper GD, Zurakowski D, Agarwal R, Bhalla T, Eisdorfer S, Huang H, Maxwell LG, Thomas JJ, Tjia I, Wilder RT, Cravero JP. Perioperative Management and In-Hospital Outcomes After Minimally Invasive Repair of Pectus Excavatum: A Multicenter Registry Report From the Society for Pediatric Anesthesia Improvement Network. Anesth Analg. 2019 Feb;128(2):315-327. doi: 10.1213/ANE.0000000000003829. PMID 30346358
- [Background] Man JY, Gurnaney HG, Dubow SR, DiMaggio TJ, Kroeplin GR, Adzick NS, Muhly WT. A retrospective comparison of thoracic epidural infusion and multimodal analgesia protocol for pain management following the minimally invasive repair of pectus excavatum. Paediatr Anaesth. 2017 Dec;27(12):1227-1234. doi: 10.1111/pan.13264. Epub 2017 Oct 24. PMID 29063665
- [Background] Gurria JP, Simpson B, Tuncel-Kara S, Bates C, McKenna E, Rogers T, Kraemer A, Platt M, Mecoli M, Garcia VF, Brown RL. Standardization of clinical care pathway leads to sustained decreased length of stay following Nuss pectus repair: A multidisciplinary quality improvement initiative. J Pediatr Surg. 2020 Dec;55(12):2690-2698. doi: 10.1016/j.jpedsurg.2020.08.009. Epub 2020 Aug 16. PMID 32972738
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068